CLINICAL TRIAL: NCT06616168
Title: Ministry of Health of Ukraine No. 2264 from 15.12.2022, Ministry of Health of Ukraine No. 310 from 08.05.2014, Ministry of Health of Ukraine No. 928 from 18.05.2023
Brief Title: Urogenital Infections in Women of Reproductive Age and the Activity of 4-Thiazolidinone Derivatives Against Pathogens
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Danylo Halytsky Lviv National Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 15.12.23, №13
Record Dates: First submitted 2024-08-28; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-08

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Penicillin G; Ceftriaxone; Doxycycline; Clindamycin; Nystatin; Amphotericin B

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Women with bacterial vaginosis (Experimental): Women with bacterial vaginosis (symptomatic or asymptomatic)
  Interventions: Diagnostic Test: Microbiological identification kits (ANAEROtest, STAPHYtest, ENTEROtest, NEFERMtest); Drug: Antibiotic therapy after the results of antibiotic sensitivity test (Mostly Oxacillin, Benzylpenicillin, Ceftriaxone, Doxycycline, Clindamycin); Combination Product: Suppositoria for vaginal microflora recovery (Giynoflor); Drug: Antifungal therapy (Mostly Fluconazole, Nystatin, Amphotericin B)
- Pregnant women (Experimental): Pregnant women with different ifections
  Interventions: Diagnostic Test: Microbiological identification kits (ANAEROtest, STAPHYtest, ENTEROtest, NEFERMtest); Drug: Antibiotic therapy after the results of antibiotic sensitivity test (Mostly Oxacillin, Benzylpenicillin, Ceftriaxone, Doxycycline, Clindamycin); Combination Product: Suppositoria for vaginal microflora recovery (Giynoflor); Drug: Antifungal therapy (Mostly Fluconazole, Nystatin, Amphotericin B)
- Women with asymptomic infections (Experimental): Women with asymptomic infections of urogenital tract
  Interventions: Diagnostic Test: Microbiological identification kits (ANAEROtest, STAPHYtest, ENTEROtest, NEFERMtest); Drug: Antibiotic therapy after the results of antibiotic sensitivity test (Mostly Oxacillin, Benzylpenicillin, Ceftriaxone, Doxycycline, Clindamycin); Combination Product: Suppositoria for vaginal microflora recovery (Giynoflor)

INTERVENTIONS:
Diagnostic Test: Microbiological identification kits (ANAEROtest, STAPHYtest, ENTEROtest, NEFERMtest) — Microbiological identification kits (ANAEROtest, STAPHYtest, ENTEROtest, NEFERMtest) produced by Erba Lachema leads to bacteria detection via biochemical features
Drug: Antibiotic therapy after the results of antibiotic sensitivity test (Mostly Oxacillin, Benzylpenicillin, Ceftriaxone, Doxycycline, Clindamycin) — Antibiotic therapy after the results of antibiotic sensitivity test. Aminoglycosides, Carbapenems, Cephalosporins, Fluoroquinolones, Oxazolidinones are used. Mostly Oxacillin, Benzylpenicillin, Ceftriaxone, Doxycycline, Clindamycin are used for the therapy.
Combination Product: Suppositoria for vaginal microflora recovery (Giynoflor) — Prescription of suppositoria for vaginal microflora recovery after antibiotic therapy. Probiotic grug includes Lactobacilli acidophillis as the main compound.
Drug: Antifungal therapy (Mostly Fluconazole, Nystatin, Amphotericin B) — Prescription of antifungal drugs. Triazoles (Fluconazole, Itraconazole, Voriconazole), Imidazoles (Ketoconazole), Nystatin and Amphotericin B are used the most
  Arms: Pregnant women; Women with bacterial vaginosis

SUMMARY:
Research concerning women pathogenic microflora during different conditions

DETAILED DESCRIPTION:
Study of microflora of different groups of women of reproductive age, determination of pathogens and their further study, samples of a newly synthesized compound on isolated pathogens

ELIGIBILITY:
Inclusion Criteria:

* urogenital infections, pregnancy

Exclusion Criteria:

* healthy microflora

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Estimation of the immune activity | 1 month
  Detection of quantities of different immune cells: lymphocytes, leukocytes, neutrophils, eosinophils
Quantities of vaginal microflore bacteria | 2 months
  Detection of quantities of vaginal microflore bacteria before and after antibiotic therapy (in TBC)

SECONDARY OUTCOMES:
Quantities of bacteria in urine | 2 months
  Detection of quantities of bacteria in urine (in TBC)

CONTACTS AND LOCATIONS:
Overall Officials: Yulian Konechnyi, Study Director — Danylo Halytsky Lviv National Medical University
Locations (1):
- Danylo Halytsky Lviv National Medical University, Lviv, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Protocol of the research — https://www.dec.gov.ua/wp-content/uploads/2023/01/knavv2022-2264.pdf